CLINICAL TRIAL: NCT07125313
Title: Effect of Yoga Training on Cardiovascular, Autonomic, Mental Health and Cognitive Parameters in Hypertensive Patients: a Randomized Controlled Clinical Trial (Hypertension and Yoga Study)
Brief Title: Effect of Yoga Training on Cardiovascular and Mental Health Parameters in Hypertensive Patients
Acronym: HY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Catarina (Other)
Responsible Party: Principal Investigator, Aline Mendes Gerage, PhD, Universidade Federal de Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HY STUDY
Record Dates: First submitted 2025-07-23; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Yoga

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YOGA (Experimental): The GY will receive an intervention involving Yoga Training (TY), which will be divided into two phases: Phase 1 (first eight weeks), which will be supervised, with three weekly sessions lasting 60 minutes, and Phase 2 (the following eight weeks), which will consist of three supervised sessions per week and the delivery of an asynchronous video lesson via a digital platform, with an incremental session of one session per week. Classes will also be 60 minutes long. The supervised sessions will take place at the UFSC CDS rehabilitation center. TY sessions will follow the following structure: breathing techniques (Pranayama), warm-up (Pavana Muktasana), physical postures in standing, sitting, and lying positions (Asanas), and relaxation (Yoganidrá). The postures will be prescribed by holding time in seconds (30 to 40 seconds), number of sets, and rest between sets. Each session will include beginner, intermediate, and advanced postures.
  Interventions: Behavioral: YOGA
- CONTROL (Other): The CG will not receive any intervention during the study and, like the GY subjects, will be instructed not to change their routines.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: YOGA — The participants randomized to the yoga group will perform 16 weeks of yoga training, three times/week for 60 minutes.
  Arms: YOGA
Behavioral: Control — Usual care
  Arms: CONTROL

SUMMARY:
The objective of this study will be to analyze the effect of 16 weeks of Yoga training on cardiovascular, autonomic, mental health, and cognitive parameters in hypertensive individuals. This is a randomized, controlled clinical trial to be conducted with adults and elderly (40 years or older), of both sexes, diagnosed with High Blood Pressure (HBP), who will be randomized into two groups: Yoga Group (YG) and Control Group (CG). The YG will undergo a Yoga training program involving breathing techniques, mobility, physical postures, relaxation, and meditation for 16 weeks. In the first eight weeks (phase 1), three supervised weekly sessions will be held. In the last eight weeks of the study (phase 2), the training will consist of three supervised weekly sessions and the delivery of an asynchronous video lesson, with the weekly frequency then increasing (from three to four sessions per week). The video lesson will be available on a digital platform. Before, after eight weeks, and after 16 weeks, cardiovascular, autonomic, mental and cognitive health parameters will be assessed. Furthermore, the biomarkers Brain-Derived Neurotrophic Factor (BDNF), serotonin, and nitric oxide will be analyzed at different assessment times of the study, as well as biochemical profile tests (glucose, total cholesterol, among others), functional capacity tests, and body composition. This project is expected to contribute to the literature by better elucidating the effects of Yoga on the cardiovascular, mental, and cognitive health of hypertensive individuals. The SPSS (21.0) statistical package will be used for data analysis. After confirming the appropriate assumptions, generalized estimating equations will be used, followed by the Bonferroni post hoc test, with a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Adults or elderly individuals
* >= 40 years
* Both sexes
* Diagnosis of hypertension controlled by up to three medications
* Who do not present high cardiovascular risk
* Who have not engaged in a physical exercise program in the six months prior to the start of the study will participate in the study.

Exclusion Criteria:

* Adherence of less than 75% of training sessions
* Diagnosis of other diseases during the study
* Adherence to another physical exercise program
* Change in the class and/or dose of antihypertensive medication during the study
* Worsening of the disease (resting systolic blood pressure (BP) > 180 mmHg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-08-11 (Estimated); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | Baseline, 8 and 16 weeks
  Clinical BP (Systolic and Diastolic) will be measured using an oscillometric device (Omron HEM 742) (OMRON Healthcare, Kyoto, Japan), according to current recommendations, while ambulatory BP will be assessed over 24 hours using a DynaMAPA device (Cardios), both in accordance with current recommendations (FEITOSA et al., 2024).

SECONDARY OUTCOMES:
Quality of life | Baseline, 8 and 16 weeks
  Quality of life will be assessed using the EuroQol 5 Dimensions 5 Levels (EQ-5D-5L) (EUROQOL, 2025; VAN ROTTERDAM, HENSLEY, HAZELTON, 2021). This questionnaire was introduced by the EuroQol Group in 2009. This questionnaire assessed quality of life and health perception, consisting of a page with an objective questionnaire and another page with a visual analog scale. The objective questionnaire is divided into five aspects: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each aspect has five levels ranging from "no problem" (1) to "extreme problem" (5), thus, higher scores denote a worse quality of life. The scale allows participants to record their overall health perception on a vertical scale, from 0 (worst health) to 100 (best health) (BAGATTINI, 2015).
Cognitive function | Baseline, 8 and 16 weeks
  Cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA) questionnaire, which comprises eight domains. The maximum score is 30 points, corresponding to the best cognitive ability (HOBSON, 2015).
Sleep Quality | Baseline, 8 and 16 weeks
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI-BR) (BERTOLAZI et al., 2011; BUYSSE, 1989). It consists of a questionnaire composed of 19 self-administered questions, followed by five questions to be answered by the bed partner, if available. This questionnaire is composed of seven domains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction (BERTOLAZI et al., 2011). Minimum: 0 points → excellent sleep and Maximum: 21 points → very poor sleep.
Depressive Symptoms | Baseline, 8 and 16 weeks
  Depressive symptoms will be assessed using the Patient Health Questionnaire-9 (PHQ-9) (APA, 2000; SANTOS et al., 2013), containing nine questions that assess the presence of symptoms of a major depressive episode, described in the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV): depressed mood, anhedonia, problems with sleep, fatigue or lack of energy, changes in appetite or weight, feelings of guilt or worthlessness, trouble concentrating, feeling sluggish or restless, and suicidal thoughts (APA, 2000). The PHQ9 assesses the frequency of symptoms in the past two weeks, assessed on a scale with the possible responses of "none of the time," "several days," "more than half the days," and "almost every day" (SANTOS et al., 2013). Values can range from 0 to 27, with higher values indicating a greater presence of depressive symptoms.
Stress | Baseline, 8 and 16 weeks
  Perceived stress will be assessed using the Perceived Stress Scale-10 (PSS-10) (SIQUEIRA REIS, FERREIRA HINO & RODRIGUEZ AÑEZ, 2010). It is an instrument that assesses the level of stress perceived by the person in recent weeks, that is, how they interpret and feel life situations as stressful. There are 10 items, each with answers from 0 to 4 points. Minimum possible: 0 points → no perceived stress and Maximum possible: 40 points → very high perceived stress. Higher values = greater perception of stress
Attention and inhibitory response capacity | Baseline, 8 and 16 weeks
  The Stroop Test will assess attention and inhibitory response capacity, calculating response time and accuracy. Better results are associated with shorter response times and fewer errors. By comparing congruent and incongruent conditions, cognitive interference and inhibitory control will be assessed (STROOP, 1935). Shorter reaction time and fewer errors → better cognitive performance and Longer reaction time and more errors → worse performance (may reflect attention difficulties, but not necessarily anxiety). There is no single universal minimum and maximum value.
Health related quality of life | Baseline, 8 and 16 weeks
  The Short Form Health Survey - 36 items (SF-36) It is a questionnaire that measures health-related quality of life in a broad way, covering physical, emotional and social aspects. Assesses 8 domains: Functional capacity, Physical aspects, Pain, General health, Vitality, Social aspects, Emotional aspects and Mental health. The SF-36 has a scoring system in which higher values indicate better, not worse, quality of life. Score for each domain: ranges from 0 to 100 0 → worst possible state 100 → best possible state Summary scores (physical and mental components) are also typically converted to this 0-100 scale (Ware; Sherboune, 1992).
Anxiety | Baseline, 8 and 16 weeks
  Hospital Anxiety and Depression Scale (HAD) is an instrument used to assess symptoms of anxiety and depression in patients. HAD-A → Anxiety Subscale (7 items) and HAD-D → Depression Subscale (7 items). Each item is scored from 0 to 3. Subscale score: Minimum: 0 points (no symptoms) and Maximum: 21 points (very severe symptoms). Higher values indicate more symptoms of anxiety or depression, depending on the subscale.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Santa Catarina, Florianópolis, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT07125313/Prot_SAP_ICF_000.pdf